CLINICAL TRIAL: NCT04753021
Title: Dose-response Relationship Between Exercise and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Collaborators: Swedish Research Council for Sport Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SwedishSchoolSHS
Record Dates: First submitted 2021-02-04; First posted 2021-02-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Mitochondrial Function; Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Progressive exercise training
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Progressively increasing training load

SUMMARY:
In this study 11 healthy volunteers will perform high intensity exercise training during 4 weeks. The exercise frequency will increase progressively during the first three weeks, followed by a fourth week with lower exercise frequency. 5 skeletal muscle biopsies will be donated throughout the study and 4 oral glucose tolerance tests will be performed after each training period.

DETAILED DESCRIPTION:
11 healthy and recreational active subjects will be recruited to the study. For inclusion and assessment of baseline physiological characteristics during cycling, a pre-test will be performed on a cycle ergometer and the submaximal and maximal response to exercise will be determined by measurement of respiratory gas exchange. The physiological response to submaximal work rate will be comprised of a series of five minutes long intervals separated with one minutes of rest with assessment of capillary blood lactate and glucose at the end of each workload. All physiological tests and training (HII) sessions will be carefully supervised by trained personnel. The intervention period will include 14 HIIT-sessions in total, all performed at the laboratory under close surveillance and careful monitoring of power output and heart rate. During HIIT sessions, VO2, CO2, blood glucose, lactate and rating of perceived exhaustion (BORG) will be measured.

Energy intake will be standardized for each subject during the day of test sessions. After each HIIT-session a recovery drink containing 1 g · kg-1 bw of carbohydrates and 0.25 g · kg-1 bw of protein will be ingested by the subjects. After HIIT sessions, subjects will be supplied with an evening meal consisting of 74 g carbohydrates, 38 g protein and 26 g fat to be consumed two hours post exercise. Subjects will thereafter remain fasted until the next morning for an oral glucose tolerance test (OGTT) and donation of a muscle biopsy.

All biopsies will be collected in fasted state in early morning following 14 hour of rest after the last HIIT-session. Biopsies will be taken from vastus lateralis in alternating leg in randomized order.

Each subject will complete four OGTTs throughout the study. Resting metabolic rate (RMR) will be measured in supine position by gas exchange measurement using mixing chamber method (Oxycon Pro) attached to a ventilated hood. Thereafter the muscle biopsy will be taken and a catheter will be inserted into the antecubital vein of the forearm. After 10 minutes of passive rest 75 mg glucose dissolved in 300 ml water will be ingested and at 0, 15, 30, 45, 60 75, 90, 105- and 120-minutes after glucose intake a venous blood sample will be taken and instantly analyzed for glucose with enzymatic method in the Biosen C-Line Clinic. Additional RMR measurements will be performed at ~40 and 115 minutes after glucose ingestion.

Mitochondria will be isolated from fresh skeletal muscle biopsies. Mitochondrial respiration and H2O2 emission will be measured using a two-channel high-resolution respirometer with an attached fluorescent probe (Oxygraph-2k, Oroboros Instruments Corporation, Innsbruck, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Endurance training of more than 5 hours a week
* regularly performing high intensity interval training (HIIT).
* Chronic medication,
* chronic diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Change in mitochondrial respiration | At baseline (before exercise training), after 1 week of training, after 2 weeks of training, after 3 weeks of training, after 4 weeks of training
  Measurement of mitochondrial oxygen consumption in isolated mitochondria from Vastus Lateralis. Respiration will be assessed using substrate combinations targeting both complex I and II. Assessment will be performed in an Oroboros oxygraph

SECONDARY OUTCOMES:
Change in glucose tolerance | At baseline (before exercise training), after 1 week of training, after 3 weeks of training, after 4 weeks of training
  Measurement of blood glucose response to 75g oral glucose
Change in oxidative stress | At baseline (before exercise training), after 1 week of training, after 2 weeks of training, after 3 weeks of training, after 4 weeks of training
  Measurement of carboylated proteins in skeletal muscle biopsies using a commercial ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Filip J Larsen, PhD, Principal Investigator — The Swedish School of Sport and Health Sciences
Locations (1):
- The Swedish School of Sport and Health Sciences (GIH), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flockhart M, Nilsson LC, Ekblom B, Larsen FJ. A Simple Model for Diagnosis of Maladaptations to Exercise Training. Sports Med Open. 2022 Nov 4;8(1):136. doi: 10.1186/s40798-022-00523-x. PMID 36333619
- [Derived] Flockhart M, Nilsson LC, Tais S, Ekblom B, Apro W, Larsen FJ. Excessive exercise training causes mitochondrial functional impairment and decreases glucose tolerance in healthy volunteers. Cell Metab. 2021 May 4;33(5):957-970.e6. doi: 10.1016/j.cmet.2021.02.017. Epub 2021 Mar 18. PMID 33740420